CLINICAL TRIAL: NCT02783976
Title: A Prospective, Non-Interventional Cohort Study of Approved Sofosbuvir-based Regimens in Patients in Mexico With Chronic Hepatitis C Virus Infection in Clinical Practice
Brief Title: Sovaldi-based Regimens in Patients in Mexico With Chronic Hepatitis C Virus Infection in Clinical Practice
Status: Completed | Type: Observational
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: GS-US-334-1685
Record Dates: First submitted 2016-05-24; First posted 2016-05-26 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: HCV Infection
MeSH Terms: conditions — Hepatitis C | interventions — Sofosbuvir

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sovaldi-based regimens: Adult patients with chronic HCV infection living in Mexico who take Sovaldi as part of routine clinical care at a participating clinical site.
  Interventions: Drug: Sovaldi

INTERVENTIONS:
Drug: Sovaldi — Sovaldi 400 mg tablets administered orally once daily
  Other Names: Sofosbuvir; GS-7977

SUMMARY:
This study will collect and evaluate information on the safety and efficacy of Sovaldi-based regimens in routine clinical practice in Mexico. The primary objective of this study is to assess the rates of serious adverse events/reactions (SAEs/SADRs) and adverse events/reactions (AEs/ADRs) in adult participants with chronic hepatitis C virus (HCV) infection treated with Sovaldi in routine clinical practice.

ELIGIBILITY:
Key Inclusion Criteria:

* HCV-infected patients living in Mexico
* Treatment with a Sovaldi-based regimen, per the approved prescribing information, as determined by the patient's treating physician

Key Exclusion Criteria:

* Concurrent participation in an HCV clinical trial (except trials not testing investigational medicinal products)
* Patients presenting a risk of not being able to be followed (eg, patients planning to move or leave the country prior to their SVR12 visit)

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with chronic HCV infection living in Mexico who take SOF as part of routine clinical care at a participating clinical site.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2016-10-28 (Actual); Primary Completion 2018-06-20 (Actual); Study Completion 2018-06-20 (Actual)

PRIMARY OUTCOMES:
Proportion of participants experiencing adverse drug reactions (ADRs), serious adverse events (SAEs), and adverse events (AEs) during the treatment period and posttreatment follow-up period | Up to Posttreatment Week 4

SECONDARY OUTCOMES:
Frequency of concurrent use of Sovaldi with amiodarone and another direct acting antiviral (DAA) or with potent intestinal P-gp inducers in routine clinical practice | Up to 24 weeks
Proportion of patients with sustained virologic response (SVR) at 12 weeks post treatment (SVR12), defined as HCV RNA < lower limit of quantification between 10 and 24 weeks post-treatment | Up to Posttreatment Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (5):
- Mexico (5):
  - Cuernavaca
  - Durango
  - Guadalajara
  - Mexico City
  - Monterrey